CLINICAL TRIAL: NCT05647824
Title: User Performance of the TV4 Blood Glucose Monitoring System
Brief Title: User Performance of the TV4 BGMS
Status: Completed | Type: Observational
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: GCA-PRO-2019-006-01
Record Dates: First submitted 2022-11-15; First posted 2022-12-13 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- All Subjects: Consists of people with Diabetes and people without Diabetes
  Interventions: Device: Capillary Testing; Device: Alternative Site Testing (AST); Device: Venous Testing

INTERVENTIONS:
Device: Capillary Testing — Testing Contour Fit BGMS with capillary blood
  Other Names: Contour Fit BGMS
Device: Alternative Site Testing (AST) — Testing Contour Fit BGMS using blood from alternative site
  Other Names: Contour Fit BGMS
Device: Venous Testing — Testing Contour Fit BGMS with venous blood
  Other Names: Contour Fit BGMS

SUMMARY:
Thunder V4 (TV4) is the code name of a blood glucose monitoring system (BGMS) consisting of a new meter and new Contour FIT test strips. This clinical trial will assess the performance (accuracy) of the TV4 meter by lay users enrolled as subjects in the study, and by health care professionals (also called study staff).

DETAILED DESCRIPTION:
The study will be conducted at three clinical sites and enroll a total of approximately 402 lay users. Ten to fifteen percent (10 - 15%) of the enrolled subjects will be naïve users (naïve to SMBG's and may include people without diabetes). At least twenty percent (20%) of subjects enrolled with diabetes will have Type 1 diabetes. At least 70% of subjects will be younger than age 65. Sites will also enroll subjects of Chinese descent.

This clinical investigation will be conducted within the US.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Ability to speak, read and understand English. Subjects must demonstrate the ability to read a paragraph from the first page of the User Guide (UG) to qualify for the study.
* Willing to complete all study procedures

Exclusion Criteria:

* Subjects without diabetes that are not naïve to Blood Glucose Monitoring System.
* Hemophilia or any other bleeding disorder
* Pregnancy (self-reported)
* Physical, visual or neurological impairments that would make the person unable to perform testing with the BGMS.
* Previous use of the Ascensia Contour Thunder V3 (TV3), or Thunder PLUS (T-PLUS), or Thunder V4 (TV4) BGMS.
* Working for a medical laboratory, hospital or another clinical setting that involves training on, or clinical use of blood glucose monitors.
* Being in this trial during or soon after xylose absorption testing (Xylose in the blood is known to cause interference). However, subjects can be enrolled as soon as 2 days after the test is performed (25 gms of oral xylose administered during this test is cleared within 480 mins or 8 hours).
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk. The reason for exclusion will be clearly documented by investigator or designee on the subject disposition form.
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.

  * Immediate family members are the subject's parents, spouse, children, and siblings, including the parent's spouse; step-children and adopted children and their spouses.
  * A competitive medical device company is a company that provides a medical device or components of a device that is related to diabetes.

For example, people who are not eligible are those who work for companies that create or manufacture the following (or a company that is in a partnership with a company that provides such devices): lancing devices, blood glucose monitoring systems, continuous glucose monitoring systems, insulin pens, or systems related to the measurement of HbA1c.

People who are eligible are those who work for companies associated with products such as wound dressings, medications or dietary products.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The following population criteria are study goals, with each site recruiting to meet these goals:
  1. Enrollment: A total of at least 402 subjects across the sites, or it can also be 134 per clinical site.
  2. At least 70% of all subjects will be younger than age 65 (across all the sites).
  3. Ten to fifteen % (10-15%) of naïve users (naïve to SMBG's and may include people without diabetes) (across all the sites).
  4. At least 20% of non-naïve users (subjects with diabetes) will have type 1 diabetes (across all the sites).
  5. Sites will also recruit subjects of Chinese descent according to the site's ability. (One or both of the subject's parents can be of Chinese descent.)
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Fingerstick Test: Obtain TV4 BGMS performance data in the hands of lay users with diabetes using fingerstick capillary blood obtained with Microlet NEXT® lancing device. | 4 weeks
  Number of glucose results falling within ±15mg/dL of laboratory method at glucose concentration <100 mg/dL and within ±15% at glucose concentrations ≥100 mg/dL

SECONDARY OUTCOMES:
Alternative Site Test (AST): Obtain TV4 BGMS performance data in the hands of lay users with diabetes using capillary blood from the palm site obtained with Microlet NEXT lancing device with the AST endcap. | 4 weeks
  Number of glucose results falling within ±15mg/dL of laboratory method at glucose concentration <100 mg/dL and within ±15% at glucose concentrations ≥100 mg/dL
Venous Blood Test: Obtain TV4 BGMS performance data using venous blood from lay users with diabetes. | 4 weeks
  Number of glucose results falling within ±15mg/dL of laboratory method at glucose concentration <100 mg/dL and within ±15% at glucose concentrations ≥100 mg/dL
Subject Questionnaire on the Usability of TV4 BGMS | 4 weeks
  Number of results with scores of 3 or higher to statements concerning instructions for use or ease of use. Scores of 3 or greater (on a scale of 0 to 5) are more favorable to usability.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Christiansen, MD, Principal Investigator — Diablo Clinical Research (DCR)
Locations (3):
- United States (3):
  - Diablo Clinical Research (DCR), Walnut Creek, California
  - Rocky Mountain Clinical Research, LLC, Idaho Falls, Idaho
  - Rainier Clinical Research Center Inc, Renton, Washington

REFERENCES:
- [Background] Protection of laboratory workers from occupationally acquired infections; approved guideline - third edition. CLSI document M29-A3. ISBN1-56238-567-4.
- [Background] Rutala W, Weber D, Healthcare Infection Control Practices Advisory Committee. Guideline for disinfection and sterilization in healthcare facilities, 2008. CDC.
- [Background] FDA, Processing/Reprocessing Medical Devices in Health Care Settings: Validation Methods and Labeling, May 2, 2011.